CLINICAL TRIAL: NCT07187687
Title: TrIal of Early Minimally Invasive Catheter Evacuation With Thrombolysis in IntraCerebral Hemorrhage (TIME-ICH): A Prospective, Multi-center, Open-label, Adaptive, Randomized Controlled Trial
Brief Title: TrIal of Early Minimally Invasive Catheter Evacuation With Thrombolysis in IntraCerebral Hemorrhage
Acronym: TIME-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIME-ICH-2025
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Intracranial Hemorrhages; ICH; brain hemorrhage; Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Minimally invasive catheter evacuation; Minimally invasive surgery; Neurosurgery; Thrombolysis; Urokinase; Medical Economic; Hospital Economics
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Hemorrhage; Cerebrovascular Disorders; Brain Diseases | interventions — Fibrinolytic Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Minimally Invasive Surgery with Thrombolysis (eMIST) plus best medical management (BMM) (Experimental): Subjects will undergo minimally invasive catheter evacuation followed by up to 10 doses of 50000U of urokinase for intracerebral hemorrhage clot resolution.
  Interventions: Procedure: Early Minimally Invasive Surgery with Thrombolysis (eMIST)
- Best medical management (BMM) (No Intervention): Subjects will receive standard of care medical management for ICH.

INTERVENTIONS:
Procedure: Early Minimally Invasive Surgery with Thrombolysis (eMIST) — Subjects will undergo minimally invasive catheter evacuation in the early stage of intracranial hemorrhage. Up to 10 doses of 50000U of urokinase will be administered through the catheter that was placed directly into the intracerebral hemorrhage.
  Arms: Early Minimally Invasive Surgery with Thrombolysis (eMIST) plus best medical management (BMM)

SUMMARY:
TIME-ICH (TrIal of early Minimally Invasive catheter Evacuation with thrombolysis in IntraCerebral Hemorrhage) is a multicenter, randomized, adaptive clinical trial comparing best medical management to early minimally invasive surgery with thrombolysis (eMIST) in the treatment of acute spontaneous supratentorial intracerebral hemorrhage.

DETAILED DESCRIPTION:
Patients presenting to the emergency department with stroke due to supratentorial, spontaneous intracerebral hemorrhage ≥20mL volume will be assessed to determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomized 1:1 using central computerized allocation to early minimally invasive surgery with thrombolysis versus best medical management. The trial is prospective, randomized, open-label, blinded endpoint (PROBE) design. Adaptive sample size re-estimation will be performed when 250 patients have completed 180 days follow-up. Clinical efficacy will be determined by demonstrating an improvement in functional outcome, as determined by a blinded-assessment of the 180-day utility-weighted modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Pre-randomization head CT demonstrating an acute, spontaneous, primary ICH;
3. ICH volume ≥ 20mL as calculated by the ABC/2 method;
4. The randomization can be completed within 8 hours after the onset of stroke symptoms (or the time last known to be well), and study intervention can reasonably be initiated within 4 hours after randomization.
5. Historical Modified Rankin Score 0 or 1;
6. Obtain informed consent from patient or legal representative.

Exclusion Criteria:

1. Infratentorial intraparenchymal hemorrhage including midbrain, pontine, or cerebellar;
2. Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, venous sinus thrombosis, mass or tumor, hemorrhagic conversion of an ischemic infarct, tumor stroke, recurrence of a recent (<1 year) ICH, as diagnosed with radiographic imaging;
3. Presence of spot sign in CT angiography;
4. Blood pressure control before randomization is ineffective, systolic blood pressure > 220 mmHg;
5. Irreversible impaired brain stem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS ≤ 4;
6. Hemorrhage with apparent midbrain extension with third nerve palsy or dilated and non-reactive pupils. Other (supranuclear) gaze abnormalities are not exclusions;
7. Intraventricular extension of the Hemorrhage is visually estimated to involve >50% of either of the lateral ventricles;
8. Any irreversible coagulopathy or known clotting disorder.
9. Platelet count < 750,000, INR > 1.4 after correction
10. Patients requiring long-term anti-coagulation that needs to be initiated < 30 days from index ICH;
11. Use of 2 or more antithrombotic drugs prior to symptom onset;
12. Patients with a mechanical heart valve;
13. Positive urine or serum pregnancy test in female subjects without documented history of surgical sterilization or is post-menopausal;
14. Urokinase allergy;
15. Any concurrent serious illness that would interfere with the outcome assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease;
16. Inability or unwillingness of patient or legal representative to give written informed consent;
17. Known life-expectancy of less than 6 months;
18. Participation in a concurrent interventional medical investigation or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional Improvement - uw-mRS | 180 days
  Functional Improvement as determined by utility-weighted modified Rankin Scale (uw-mRS) which is assigned to seven levels: 1.0, 0.91, 0.76, 0.65, 0.33, 0.0, and 0.0 (with higher scores indicating a better outcome, according to patients' assessment) at 180-days.

SECONDARY OUTCOMES:
Functional Improvement - uw-mRS | 7 days, 14 days (discharge), 30 days and 90 days
  Functional Improvement as determined by utility-weighted modified Rankin Scale (uw-mRS) which is assigned to seven levels: 1.0, 0.91, 0.76, 0.65, 0.33, 0.0, and 0.0 (with higher scores indicating a better outcome, according to patients' assessment) at 7 days, 14 days/discharge, 30 days and 90 days.
Functional Improvement - good functional outcome | 7 days, 14 days (discharge), 30 days, 90 days and 180 days
  Good functional outcome as determined by modified Rankin Scale (mRS) 0-3 at 7 days, 14 days/discharge, 30 days, 90 days and 180 days
Mortality | 180 days
  Mortality at 180 days.
Clot Removal - Amount of Residual Blood | 36 hours, 7 days and 14 days (discharge)
  Clot Removal will be assessed by the amount of residual blood at 36 hours, 7 days and 14 days/discharge.
Health-related quality of life - EQ-5D-5L | 14 days (discharge), 30 days, 90 days and 180 days
  Health-related quality of life will be assessed by EuroQol five-dimension, five-level (EQ-5D-5L) which consists of two parts, a short descriptive system questionnaire and a visual analogue scale (EQ VAS) at 7 days, 14 days/discharge, 30 days, 90 days and 180 days.
Activities of Daily Living - Barthel Index | 14 days (discharge), 30 days, 90 days and 180 days
  Activities of Daily Living will be assessed by Barthel Index at 14 days/discharge, 30 days, 90 days and 180 days.

OTHER OUTCOMES:
Safety - All Cause Mortality | 30 days
  Safety will be assessed by mortality from all causes at 30 days.
Safety - Procedure-Related Mortality | 7 days
  Safety will be assessed by procedure-related mortality at 7 days.
Safety - Bacterial intracranial infection | 30 days
  Safety will be assessed by brain bacterial infection events at 30 days.
Safety - Symptomatic Brain Bleeding Within 72 Hours After Last Dose | 72 hours after last dose
  Safety will be assessed by adjudicated symptomatic brain bleeding events within 30 days.
Economic | 14 days (discharge), 30 days, 90 days and 180 days.
  Economic differential as determined by quantification of the cost per quality-adjusted life-years (QALY) gained through eMIST.

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - Guangdong Provincial People's Hospital, Guangdong, Yuexiu
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Beijing Daxing District People's Hospital, Beijing
  - Beijing Fengtai You'anmen Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Changsha Central Hospital, Changsha
  - Changzhi Medical College Affiliated Heji Hospital, Changzhi
  - Chifeng Municipal Hospital, Chifeng
  - Chongqing Emergency Medical Service, Chongqing
  - First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jinan City People's Hospital, Jinan
  - Jinan Hospital of Xuanwu Hospital, Capital Medical University, Jinan
  - The First People Hospital of Yunnan Province, Kunming
  - Tibet People's Hospital, Lhasa
  - Liaocheng Brain Hospital, Liaocheng
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Hospital of Nantong University, Nantong
  - Center Hospital of Nanyang, Nanyang
  - Third People's Hospital of Hainan Province, Sanya
  - Shanghai Fourth People's Hospital Affiliated to Tongji University, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Suining Central Hospital, Sichuan
  - Central People's Hospital of Siping City, Siping
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an
  - Tianjin Huanhu Hospital, Tianjin
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Yanan Medical College of Yanan University, Yan’an
  - Henan Provincial People's Hospital, Zhengzhou
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The Fourth People's Hospital of Zigong City, Zigong

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other parties to maximize the usefulness of the collected research data. Data can be requested from the principal investigators with a detailed description of the objectives and methods of the study for which the data is intended. Data will be made available for this purpose at least 18 months after the publication of the main report.
Supporting Information: Study Protocol, SAP
Time Frame: At least 18 months after the publication of the main report.
Access Criteria: Written proposals will be assessed by TIME-ICH investigators for appropriateness of use, and a data sharing agreement in accordance with China regulations will be put in place before data is shared.